CLINICAL TRIAL: NCT06758219
Title: Validity and Reliability of the Turkish Form of the Knowledge Assessment Scales for Dementia and Urinary Incontinence
Status: Recruiting | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Atahan TURHAN, Dr. Lecturer, Kirsehir Ahi Evran Universitesi
Other Study IDs: KAEU-T.ATAHAN-007
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-11

CONDITIONS: Urinary Incontinence in Old Age; Dementia
Keywords: Urinary Incontinence; Dementia; Validity; Reliability
MeSH Terms: conditions — Dementia; Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group
  Interventions: Other: There is no intervention in the study.

INTERVENTIONS:
Other: There is no intervention in the study. — There is no intervention in the study.

SUMMARY:
The primary aim of the study was to determine the Turkish version of the "Validity and Reliability of the Knowledge Assessment Scales for Dementia and Urinary Incontinence in Community Older People". The secondary aim of the study was to measure the knowledge level of dementia and urinary incontinence in the community-living elderly population.

ELIGIBILITY:
Inclusion Criteria:

1. Being 55 years of age or older
2. Knowing how to read and write
3. Being willing to participate in the study

Exclusion Criteria:

1. Having any chronic illness that would prevent urinary retention and dementia level

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be conducted at Kırşehir Ahi Evran University Physical Therapy and Rehabilitation Center. All patient relatives and hospital staff who meet the inclusion criteria will be included in the study. These participants will be reached through face-to-face communication or online methods (sms, e-mail), and a list of participants will be prepared and evaluations will be made.
Sampling Method: Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2024-12-08 (Actual); Primary Completion 2025-07-10 (Estimated); Study Completion 2025-08-10 (Estimated)

PRIMARY OUTCOMES:
Knowledge Assessment Scales for Dementia and Urinary Incontinence in Community Older People | 20 weeks
  The scale was developed by Hui Sun et al. to assess the level of knowledge about dementia and urinary incontinence among elderly individuals living in the community. The original language of the scale is Chinese and was translated into English by the researchers. The two knowledge assessment scales for dementia and urinary incontinence consist of 12 and 8 items, respectively. The model fit indicators of both met the criteria of confirmatory factor analysis. Cronbach'sα was 0.82 and 0.70, respectively. The completion rate and completion time of the two scales were 83.51% and 4.22±1.90 minutes.

SECONDARY OUTCOMES:
International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF) | 20 weeks
  The severity of incontinence and its impact on the quality of life of the participants will be assessed with the ICIQ-SF. The ICIQ-SF consists of 6 items that question the type and frequency of urinary incontinence and the impact of incontinence on the individual's quality of life. The total score that can be obtained from the scale varies between 0-21. An increase in the total score indicates an increase in the severity of incontinence.
Incontinence Quality of Life Questionnaire (I-QOL) | 20 weeks
  The participants' quality of life will be assessed with the I-QOL, which was specifically developed for urinary incontinence. The I-QOL is a scale consisting of 22 items and 3 subgroups that questions thoughts such as anxiety and depression that develop due to incontinence and the reflection of these thoughts on life. The total score that can be obtained from the scale varies between 0-100, and higher scores indicate better quality of life.
Standardize Mini Mental State (SMMS) | 20 weeks
  SMMS will be used to assess the cognitive status of the participants. SMMS is a scale consisting of 11 items and 5 subgroups that measure cognitive functions. The total score that can be obtained from the scale varies between 0-30, and it is recommended that those who score 24 and below be evaluated for dementia.
Lawton-Brody Instrumental Activities of Daily Living Scale (IADL) | 20 weeks
  The independence of the participants in their daily living activities will be assessed with the IADL. The IADL is a scale consisting of 8 items that assess instrumental daily living activities. The total score that can be obtained from the scale varies between 0-24, and an increase in the score indicates an increase in the level of independence.

CONTACTS AND LOCATIONS:
Locations (1):
- Kirsehir Ahi Evran University Physical Therapy and Rehabilitation Center, Kırşehir, Merkez, Turkey (Türkiye)